CLINICAL TRIAL: NCT02146313
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety, Tolerability, and Pharmacokinetics of DMUC4064A Administered Intravenously to Patients With Platinum-Resistant Ovarian Cancer or Unresectable Pancreatic Cancer
Brief Title: A Study Evaluating the Safety and Pharmacokinetics of DMUC4064A in Participants With Platinum-Resistant Ovarian Cancer or Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29213
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Neoplasms; Ovarian Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose-escalation Cohort (Experimental): DMUC4064A will be administered to participants at a starting dose of 1.0 milligram per kilogram (mg/kg) by IV infusion q3w and would be monitored for DLTs for 21 days after first infusion of Cycle 1 (cycle length=21 days).
  Interventions: Drug: DMUC4064A
- Platinum-resistant Ovarian Cancer Dose-expansion Cohort (Experimental): Platinum-resistant Ovarian Cancer participants will be administered with the identified RP2D during the Dose-escalation of DMUC4064A q3w IV for up to until disease progression or death, whichever occurs first.
  Interventions: Drug: DMUC4064A
- Unresectable Pancreatic Cancer Dose-expansion Cohort (Experimental): Unresectable pancreatic cancer participants will be administered with the identified RP2D during the dose-escalation of DMUC4064A q3w IV for up to until disease progression or death, whichever occurs first.
  Interventions: Drug: DMUC4064A

INTERVENTIONS:
Drug: DMUC4064A — Participants will receive escalated DMUC4064A dose or RP2D, as a single agent by intravenous (IV) infusion q3w on Day 1 of each cycle (21 days).

SUMMARY:
This is a Phase 1, multicenter, open-label, dose-escalation study of DMUC4064A administered by intravenous (IV) infusion every three weeks (q3w) to cancer participants. The study will employ a traditional 3 + 3 dose escalation design to determine the maximum tolerated dose (MTD) of DMUC4064A against platinum-resistant ovarian cancer. Once a q3w recommended Phase 2 dose (RP2D) is identified, two expansion cohorts (one in platinum-resistant ovarian cancer and another in unresectable pancreatic cancer) may be evaluated to further characterize the safety and activity in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Measurable disease is defined as at least one bi-dimensionally measurable non-lymph node lesion greater than or equal to (>/=) 1 centimeter (cm) on long access diameter on computed tomography (CT) or magnetic resonance imaging (MRI) scan or at least one bi-dimensionally measurable lymph node measuring >/=1.5 cm on short access diameter on CT or MRI scan
* Adequate hematologic, kidney and liver function
* Highly effective contraception as defined by the protocol Participants with Ovarian Cancer
* Histological documentation of epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
* Documentation of mucin 16 (MUC16) expression by either serum carcinoma antigen 125 (CA125) >=2 x Upper limit of normal (ULN) or by immunohistochemistry [IHC] by central review
* Disease that has progressed or relapsed during or within 6 months after the most recent treatment with a platinum-containing chemotherapy regimen
* Progression or relapse from prior platinum-based chemotherapy must be documented radiographically by RECISTv1.1 criteria

For ovarian cancer dose expansion cohorts only:

* Not more than two prior chemotherapy regimens for the treatment of platinum-resistant ovarian cancer

Participants with Pancreatic Cancer:

* Histologic documentation of incurable, locally advanced, or metastatic pancreatic ductal adenocarcinoma consisting of unresectable pancreatic ductal adenocarcinoma (i.e., participants who are not considered eligible for surgical resection with curative intent), including recurrence of previously resected disease
* Documented MUC16 expression from archival or fresh tissue by IHC central review
* Participants for whom no further standard of care therapy exists, must have received standard of care chemotherapy in the adjuvant or advanced/metastatic setting
* No more than two prior chemotherapy regimens administered for the treatment of pancreatic cancer in the adjuvant or advanced/metastatic setting

Exclusion Criteria:

* Anti-tumor therapy, including chemotherapy, biologic, experimental, or hormonal therapy within 4 weeks prior to Day 1
* Prior treatment with MUC16 targeted therapy (e.g., oregovomab [OvaRex] or abagovomab) including DMUC5754A
* Prior treatment with a monomethyl auristatin E (MMAE)-containing antibody-drug conjugate (ADC)
* Palliative radiation to bone metastases within 2 weeks prior to Day 1
* Prior radiation to lung fields
* Major surgical procedure within 4 weeks prior to Day 1
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (including human immunodeficiency virus [HIV] and atypical mycobacterial disease but excluding fungal infections of the nail beds) at study enrollment or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 4 weeks prior to Cycle 1, Day 1
* Evidence of significant uncontrolled concomitant diseases, such as ocular toxicities, diabetes, cardiovascular disease; nervous system, renal, hepatic, endocrine, or gastrointestinal disorders; autoimmune disease, or a serious non-healing wound or fracture
* Clinically significant pulmonary symptoms and signs, any active pulmonary or respiratory infection at enrollment, pulmonary infiltrates on screening CT scan of the chest that are associated with symptoms (including dyspnea), resting or exercise arterial oxygen saturation (SpO2) less than (<) 90 percent (%), requirement for supplementary oxygen at rest or exercise (either continuously or intermittently), moderate (40%-60% predicted) or severe (<40% predicted) decreased diffusing capacity for carbon monoxide (DLCO) or mild (>60% </= lower limit of normal [LLN]% predicted) decrease with clinically significant symptoms
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix, squamous carcinoma of the skin, adequately controlled limited basal cell skin cancer, or synchronous primary endometrial cancer or prior primary endometrial cancer if protocol criteria are met
* Untreated or active central nervous system (CNS) metastases. Participants with a history of treated CNS metastases may be eligible
* Current Grade greater than (>) 1 toxicity (except alopecia and anorexia) from prior therapy or Grade >1 neuropathy from any cause
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Pregnancy or breastfeeding
* Inability to comply with study and follow-up procedures
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the participants at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06-22 (Actual); Primary Completion 2018-06-18 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 21 of Cycle 1 (Cycle length[CL]= 21 days)
Maximum Tolerated Dose of DMUC4064A | Day 1 up to Day 21 of Cycle 1 (CL=21 days)
Recommended Part II Dose of DMUC4064A | Baseline up to safety-follow up (approximately 3.5 years)
Percentage of Participants with Adverse Events (AEs) or Serious Adverse Events (SAEs) | Baseline up to safety-follow up (approximately 3.5 years)

SECONDARY OUTCOMES:
Percentage of Participants with Anti-DMUC4064A Antibodies | Pre-dose (0 hour[H];post infusion (infusion=90 minutes for C1; 30 minutes for C2 and beyond) on Day 1 of Cycle (C) 1-4; at study completion or early termination (approximately 3.5 years (CL=21 days)
Pharmacokinetic (PK) Profile of DMUC4064A in Participants With Platinum-Resistant Ovarian Cancer or Unresectable Pancreatic Cancer | Days 1,2,4,8,11,15 of C1;Days 8,15 of C2-4; at study completion or early termination (approximately 3.5 years)
Percentage of Participants With Objective Response as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | At baseline and even numbered cycles and at study termination (approximately 3.5 years) (CL=21 days)
Duration of Objective Response | At baseline and even numbered cycles and at study termination (approximately 3.5 years) (CL=21 days)
Progression-free Survival (PFS) as Assessed by RECIST v1.1 | Day 1 of C1 until disease progression or death within 30 days of the last study drug administration, whichever occurs first (approximately 3.5 years) (CL=21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (7):
  - Florida Cancer Specialists - Sarasota (North Catttlemen Rd), Sarasota, Florida
  - Massachusetts General Hospital., Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Hackensack Univ Med Ctr, Hackensack, New Jersey
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - University of Wisconsin, Madison, Wisconsin